CLINICAL TRIAL: NCT05379894
Title: Modified Supine vs Prone Position Percutaneous Nephrolithotripsy (PNL )in Management of Complex Renal Stones, A Randomized Comparative Study
Brief Title: Modified Supine vs Prone Position Pnl
Status: Recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Mohamed El Taher, Assistant Lecturer, Assiut University
Other Study IDs: Kidney stones , PNL
Record Dates: First submitted 2022-05-10; First posted 2022-05-18 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group (1 ) Modified Supine: Modified Supine position PNL
  Interventions: Procedure: Percutaneous nephrolithotripsy
- group (2) prone: Prone position PNL
  Interventions: Procedure: Percutaneous nephrolithotripsy

INTERVENTIONS:
Procedure: Percutaneous nephrolithotripsy — Extraction of kidney stones through skin using nephroscope
  Other Names: PNL

SUMMARY:
perform a comparative randomized trial comparing the efficacy and safety of percutaneous nephrolithotomy (PCNL) in the prone and modified supine positions in management of complex renal stones

DETAILED DESCRIPTION:
since the first successful removal of a renal calculus via a nephrostomy tract in 1976, percutaneous nephrolithotomy (PCNL) has become the preferred method of treating patients with large or complex stones.1 Traditionally, PCNL has been performed in the prone position, which allows a wide field for kidney puncture, avoids abdominal visceral injuries, and makes the puncture pathway short and straight. Multiple routes of access and the interoperative use of C-arm fluoroscopy X-ray machines may contribute to the vertical positioning of the puncture. This position provides posterior access to the collecting system, which theoretically enables the surgeon to puncture a posterior calyx through Braudel's avascular renal plane without significant parenchymal bleeding and peritoneal perforation. However, the prone position also has some disadvantages. For example, abdominal pressure decreases end expiratory lung volume and lung capacity, reducing the ability of patients to tolerate prolonged surgery, contraindicating the prone position in morbidly obese patients and individuals with some respiratory diseases.

An alternative position for PCNL consists of the modified supine position, in which patients are placed in a supine position with a water bag or specially designed cushion under the flank. The modified supine position has several advantages. Due to greater comfort, the position has a low impact on a patient's blood circulation and respiratory system. This position makes it easier for the anesthetist to monitor the patient, and it may decrease the use of anesthetics. For high-risk patients, the modified supine position can be changed to facilitate endotracheal intubation anesthesia whenever needed. Moreover, the smaller angle between the horizon and the operating channel improves the removal of crushed stones. This position also facilitates simultaneous ureteroscopy access when necessary, allowing for the combination of PCNL and the ureteroscopy in the management of complex stone diseases. The major disadvantage of the modified supine position is that the kidney is more easily pushed forward by the puncture needle and the fascial dilators, leading to the establishment of a deeper channel.

It remains unclear whether the traditional prone position or the modified supine position is optimal for PCNL. The prone position has been associated with reduced operation times and higher stone clearance rates, whereas the supine position has been associated with greater safety. The Valdivia position improved by Galdakao enables the use of flexible ureteroscopy and an ureteroscopy to treat ureteral and kidney stones at the same time, whereas the Valdivia position improved by Barts often requires X-rays combined with ultrasound for determining the puncture site, and the puncture route is longer. the investigators did not utilize the Galdakao improvement of the Valdivia position since flexible ureteroscopy was too expensive for routine use. Therefore, the investigators compared the efficacy and safety of PCNL in the traditional prone and modified supine positions.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:
* Grade II - A solitary stone in the upper pole with simple anatomy or multiple stones in a patient with simple anatomy or any solitary stone in a patient with abnormal anatomy
* Grade III - Multiple stones in a patient with abnormal anatomy or, stones in a calyceal diverticulum or partial staghorn calculus
* Grade IV - Staghorn calculus or any stone in a patient with spina bifida or spinal injury.

Exclusion Criteria:

* · Pediatric group
* Grade I - A solitary stone in the mid/lower pole with simple anatomy or a solitary stone in the pelvis with simple anatomy

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients with renal stones candidate for operation
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
comparing the efficacy and safety of percutaneous nephrolithotomy (PCNL) in the prone and modified supine position | 4 years
  number of participants completely stone-free
comparing the efficacy and safety of percutaneous nephrolithotomy (PCNL) in the prone and modified supine position | 4 years
  measure amount of blood loss
comparing the efficacy and safety of percutaneous nephrolithotomy (PCNL) in the prone and modified supine position | 4 years
  measure of Time of operation

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit facility of medicine, Asyut, Assuit, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gokce MI, Ibis A, Sanci A, Akinci A, Bagci U, Agaoglu EA, Suer E, Gulpinar O. Comparison of supine and prone positions for percutaneous nephrolithotomy in treatment of staghorn stones. Urolithiasis. 2017 Dec;45(6):603-608. doi: 10.1007/s00240-017-0977-y. Epub 2017 Mar 29. PMID 28357451
- [Result] McCahy P, Rzetelski-West K, Gleeson J. Complete stone clearance using a modified supine position: initial experience and comparison with prone percutaneous nephrolithotomy. J Endourol. 2013 Jun;27(6):705-9. doi: 10.1089/end.2012.0650. Epub 2013 Mar 18. PMID 23363334